CLINICAL TRIAL: NCT04464616
Title: The Effect of Adding Dexmedetomidine or Dexamethasone to Bupivacaine-Fentanyl Mixture in Spinal Anesthesia for Cesarean Section
Brief Title: Adding Different Additives to Bupivacaine-fentanyl Mixture in Spinal Anesthesia for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: spinal additives in CS
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): spinal anesthesia with 10 mg hyperbaric bupivacaine 5% (2 ml) + 25 μg fentanyl (0.5 ml) + normal saline (0.5 ml).
  Interventions: Procedure: spinal anaesthesia
- Dexmedetomidine group): (Experimental): spinal anesthesia with 10 mg hyperbaric bupivacaine 5% (2 ml) + 25 μg fentanyl (0.5 ml) + 5 μg dexmedetomidine in a volume of (0.5 ml).
  Interventions: Procedure: spinal anaesthesia
- Dexamethasone group (Experimental): spinal anaesthesia with 10 mg hyperbaric bupivacaine 5% (2 ml) + 25 μg fentanyl (0.5 ml) + 2 mg dexamethasone in a volume of 0.5 ml).
  Interventions: Procedure: spinal anaesthesia

INTERVENTIONS:
Procedure: spinal anaesthesia — spinal anaesthesia will be performed with the patient in sitting position at the L3-L4 or L4-L5 interspaces with a 25 or 27 G spinal tip needle with the study drug in the total volume of 3 ml.
  Other Names: intrathecal anaesthesia

SUMMARY:
Spinal anesthesia is widely used in cesarean section, but it is associated with high incidence of side effects. To reduce the occurrence of side effects, intrathecal adjuvant was recommended to use in spinal anesthesia, with the aim in reducing the dose of intrathecal local anesthetic, which can subsequently decrease the incidence of spinal-induced side effects and prolong postoperative analgesia.

DETAILED DESCRIPTION:
Spinal anesthesia is widely used in cesarean section, but it is associated with high incidence of side effects. To reduce the occurrence of side effects, intrathecal adjuvant was recommended to use in spinal anesthesia, with the aim in reducing the dose of intrathecal local anesthetic, which can subsequently decrease the incidence of spinal-induced side effects and prolong postoperative analgesia.Many augmentation strategies for intrathecal analgesia have been proposed. A meta-analysis by Popping et al. concluded that the concomitant use of an opioid such as fentanyl intrathecally allows the reduction in the dose of local anesthetic, while augmenting its analgesic potency thereby decreasing its adverse effects.

Dexamethasone relieves pain through reducing inflammation and blocking of nociceptive C- fibers transmission and by suppressing neural ectopic discharge. Post-operative analgesic effectiveness and duration was prolonged when dexamethasone was used as an adjunct for peripheral nerve blocks. Recent studies reported no complications associated with intrathecal dexamethasone.

Dexmedetomidine (DEX) is a potent, selective α2 adrenergic agonist and when given intrathecally, it exerts its analgesic effect via stimulating spinal α2 receptors. Wu et al., in their meta-analysis showed that addition of intrathecal DEX significantly increased the duration of postoperative analgesia and reduced analgesic consumption. The increase in duration of postoperative analgesia is dose dependent but with increase in the incidence of bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* 90 parturient
* the statue of American Society of Anesthesiologists' physical class II
* prepared for an elective cesarean section.

Exclusion Criteria:

* BMI > 35kg/m2
* gestational age < 28 weeks
* diabetes or gestational diabetes
* hypertension or pre-eclampsia
* contraindications to spinal anesthesia
* height less than 160 Cm
* history of psychiatric disease
* taking α-receptor antagonist drugs -a history of allergy to the study drugs-
* excessive hemorrhage needing transfusion.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
time for the first request of rescue analgesia | postoperative first day
  time for the first request of rescue morphine analgesia at dose of 3 mg

SECONDARY OUTCOMES:
Numerical Rating Scale | postoperative first day
  Numerical Rating Scale (NRS) for pain that ranged from (0 = no pain) to (10 = intolerable pain). If score is >3 will need analgesia in the form of morphine 3 mg will be given till NRS decreases to ≤3. NRS will be assessed and recorded immediately postoperative, 2, 4, 8, 12, 18, 24 h after the operation, by an anesthesiologist, who is blinded to the study groups.
Maternal satisfaction | postoperative first day
  Maternal satisfaction will be evaluated on a 0-3 score (0 = poor, 1 = fair, 2 = good, and 3 = excellent).
Neonatal outcome | time of delivery of fetus
  Neonatal outcome will be assessed in terms of Apgar score.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt